CLINICAL TRIAL: NCT04144036
Title: A Phase I Trial of Neihulizumab for the Upfront Treatment of Standard-Risk, Ann Arbor Scoring 1-2 Acute Graft vs Host Disease
Brief Title: Neihulizumab for Standard-Risk Acute Graft Versus Host Disease (GVHD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sameem M. Abedin, MD (Other)
Responsible Party: Sponsor-Investigator, Sameem M. Abedin, MD, Assistant Professor, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO36517
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Graft-versus-host Disease
Keywords: Graft-versus-host disease; Neihulizumab
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Neihulizumab Dose Escalation, 3 mg/kg (Experimental): Initial dose will be 6 mg weekly and the highest dose administered will be 9 mg weekly. Patients will be entered sequentially to each dose level. If 0 of the first 3 patients at that level has a DLT, new patients may be entered at the next higher dose level. If 1 of 3 patients has a DLT, up to 3 more patients are to be treated at that same dose level. If 0 of the additional 3 patients at that dose level has a DLT, new patients may be entered at the next higher dose level. If 1 or more of the additional 3 patients experience a DLT, 0 patients are to be started at that dose level and the preceding dose is the MTD. If 2 of 3 of the dosed patients has a DLT on the first dose level, the drug will be administered at a lower dose, 3 mg weekly. If 0 of 3 patients has a DLT at the highest dose level, an additional 3 patients will be enrolled to ensure that 6 patients are treated at the MTD. The MTD is the highest dose level at which no more than 1 of 6 treated patients, experiences a DLT.
  Interventions: Biological: Neihulizumab, 3 mg/kg
- Neihulizumab Dose Escalation, 6 mg/kg (Experimental): Initial dose will be 6 mg weekly and the highest dose administered will be 9 mg weekly. Patients will be entered sequentially to each dose level. If 0 of the first 3 patients at that level has a DLT, new patients may be entered at the next higher dose level. If 1 of 3 patients has a DLT, up to 3 more patients are to be treated at that same dose level. If 0 of the additional 3 patients at that dose level has a DLT, new patients may be entered at the next higher dose level. If 1 or more of the additional 3 patients experience a DLT, 0 patients are to be started at that dose level and the preceding dose is the MTD. If 2 of 3 of the dosed patients has a DLT on the first dose level, the drug will be administered at a lower dose, 3 mg weekly. If 0 of 3 patients has a DLT at the highest dose level, an additional 3 patients will be enrolled to ensure that 6 patients are treated at the MTD. The MTD is the highest dose level at which no more than 1 of 6 treated patients, experiences a DLT.
  Interventions: Drug: Neihulizumab, 6 mg/kg
- Neihulizumab Dose Escalation, 9 mg/kg (Experimental): Initial dose will be 6 mg weekly and the highest dose administered will be 9 mg weekly. Patients will be entered sequentially to each dose level. If 0 of the first 3 patients at that level has a DLT, new patients may be entered at the next higher dose level. If 1 of 3 patients has a DLT, up to 3 more patients are to be treated at that same dose level. If 0 of the additional 3 patients at that dose level has a DLT, new patients may be entered at the next higher dose level. If 1 or more of the additional 3 patients experience a DLT, 0 patients are to be started at that dose level and the preceding dose is the MTD. If 2 of 3 of the dosed patients has a DLT on the first dose level, the drug will be administered at a lower dose, 3 mg weekly. If 0 of 3 patients has a DLT at the highest dose level, an additional 3 patients will be enrolled to ensure that 6 patients are treated at the MTD. The MTD is the highest dose level at which no more than 1 of 6 treated patients, experiences a DLT.
  Interventions: Drug: Neihulizumab, 9 mg/kg
- Neihulizumab Dose Expansion (Experimental): Upon determination of the maximum-tolerated dose, an expansion cohort of 4-7 patients will be enrolled so that a total of 10 patients are enrolled at the potential Phase II dose. This will be done to preliminarily assess efficacy.
  Interventions: Drug: Neihulizumab

INTERVENTIONS:
Biological: Neihulizumab, 3 mg/kg — The doses for the 3 + 3 design (dose escalation phase) are listed in the arm description. The dose-expansion phase will use the maximum-tolerated dose.
  Other Names: AbGn 168; AbGn 168H
  Arms: Neihulizumab Dose Escalation, 3 mg/kg
Drug: Neihulizumab, 6 mg/kg — The doses for the 3 + 3 design (dose escalation phase) are listed in the arm description. The dose-expansion phase will use the maximum-tolerated dose.
  Other Names: AbGn 168; AbGn 168H
  Arms: Neihulizumab Dose Escalation, 6 mg/kg
Drug: Neihulizumab, 9 mg/kg — The doses for the 3 + 3 design (dose escalation phase) are listed in the arm description. The dose-expansion phase will use the maximum-tolerated dose.
  Other Names: AbGn 168; AbGn 168H
  Arms: Neihulizumab Dose Escalation, 9 mg/kg
Drug: Neihulizumab — This arm will receive the Maximum Tolerated Dose determined in the Drug Escalation phase.
  Other Names: AbGn 168; AbGn 168H
  Arms: Neihulizumab Dose Expansion

SUMMARY:
This is a single-center Phase I study to determine the maximum tolerated dose and safety of Neihulizumab for the treatment of Minnesota standard-risk aGVHD. Patients undergoing allogeneic transplant with either a myeloablative or non-myeloablative conditioning regimen, and recipients of all donor sources will be enrolled to this trial.

DETAILED DESCRIPTION:
Eligible patients will receive Neihulizumab weekly, for up to four doses. Responding patients, and patients with stable disease should receive all four weekly doses. Patients with skin only disease that clinically progresses by one stage (e.g, from stage 2 to stage 3), but remains less than stage 4, will receive a minimum two doses of Neihulizumab. At 72 hours after the second dose, non-responding patients will be withdrawn from the study. Responding patients should remain on study and receive four total doses. Patients with lower GI GVHD that progresses by at least one stage at 4 or more days after first dose will be withdrawn from the study. All patients receiving at least 1 dose of Neihulizumab will be evaluated for dose-limiting toxicities (DLTs) and adverse events.

Dose-escalation will be conducted according to a 3+3 design. The initial dose of Neihulizumab will be 6 mg/kg weekly (Dose level 1), and the highest dose administered will be 9 mg/kg weekly (Dose level 2). The DLT observation period will be 28 days. Patients will be entered sequentially to each dose level. For each dose level, if none of the first 3 patients at that level experiences a DLT, new patients may be entered at the next higher dose level. If 1 of 3 patients experiences a DLT, up to 3 more patients are to be treated at that same dose level. If none of the additional 3 patients at that dose level experiences a DLT, new patients may be entered at the next higher dose level. However, if 1 or more of the additional 3 patients experience a DLT, then no further patients are to be started at that dose level and the preceding dose is the maximum-tolerated dose (MTD). If 2 of 3 of the initially dosed patients experience a DLT on the first dose level, Neihulizumab will be administered at a lower dose, 3mg/kg weekly (Dose level -1). Finally, if 0 of 3 patients experience DLT at the highest dose level, an additional 3 patients will be enrolled to ensure that 6 patients are treated at the MTD. The MTD will be defined as the highest dose level at which no more than 1 of 6 treated patients, experiences a DLT.

Upon determination of MTD, an expansion cohort of 4-7 patients will be enrolled so that a total of 10 patients are enrolled at the potential Phase II dose. This will be done to preliminarily assess efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years.
2. Recipients of myeloablative and non-myeloablative, reduced-intensity conditioning allogeneic transplants.
3. Recipients of all donor sources, including sibling, unrelated donor, human leukocyte antigen (HLA) -haploidentical, and HLA-mismatched donors.
4. Patients must have initial presentation of standard-risk aGVHD according to refined Minnesota Criteria. Standard-risk aGVHD is defined as follows:

   Single organ involvement:
   * Stage 1-3 skin
   * Stage 1 upper GI
   * Stage 1-2 lower GI

   Multiple organ involvement:
   * Stage 1-3 skin plus stage 1 upper GI
   * Stage 1-3 skin plus stage 1 lower GI
   * Stage 1-3 skin plus stage 1 lower GI plus stage 1 upper GI
   * Stage 1-3 skin plus stage 1-4 liver
   * Stage 1 lower GI plus stage 1 upper GI
5. Patients must not have received prior systemic immune suppressive therapy for the treatment of active aGVHD (topical steroids and budesonide are permitted).
6. Biopsy confirmation of GVHD is not required, but encouraged.
7. Female patients must meet one of the following:

   * Postmenopausal for at least one year before the screening visit, or
   * Surgically sterile (i.e. undergone a hysterectomy or bilateral oophorectomy), or
   * If subject is of childbearing potential (defined as not satisfying either of the above two criteria), agree to practice two acceptable methods of contraception (combination methods requires use of two of the following: diaphragm with spermicide, cervical cap with spermicide, contraceptive sponge, male or female condom, hormonal contraceptive) from the time of signing of the informed consent form through 90 days after the last dose of study agent, AND o Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptom-thermal, post ovulation methods] and withdrawal are not acceptable contraception methods).
8. Male patients, even if surgically sterilized (i.e., status post vasectomy), must agree to one of the following:

   * Practice effective barrier contraception during the entire study period and through 60 calendar days after the last dose of study agent, OR
   * Must also adhere to the guidelines of any study-specific pregnancy prevention program, if applicable, OR o Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptom-thermal, post ovulation methods] and withdrawal are not acceptable methods of contraception.)
9. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Relapse of disease which was the primary indication for transplant.
2. Uncontrolled infections not responding to antimicrobial therapy.
3. Active and uncontrolled human immunodeficiency virus (HIV), or chronic Hepatitis B, or Hepatitis C.
4. Tuberculosis, history of tuberculosis or a known positive Quantiferon test.
5. Liver dysfunction not attributable to aGVHD evidenced by a Total Bilirubin ≥ 2 x upper limit of normal (ULN).
6. Creatinine clearance < 40 mL/min calculated by Cockcroft-Gault equation.
7. Intestinal obstruction within three days of enrollment.
8. Life expectancy of less than 28 days, or Eastern Cooperative Oncology Group (ECOG) performance status of 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose. | Up to 28 days
  The maximum-tolerated dose will be defined as the highest dose level at which no more than one of six treated patients, experiences a dose-limiting toxicity.

SECONDARY OUTCOMES:
Treatment response: Complete response | Day 28
  This outcome measures the number of patients with complete response. A complete response is GVHD that fully resolves at all sites. This will be determined by assessment of aGVHD response. Acute GVHD will be assessed by Mount Sinai Acute GVHD International Consortium (MAGIC) algorithm.
Treatment response: Partial response | Day 28
  This outcome measures the number of patients with partial response. A partial response is GVHD that improves by at least one stage at one site, without worsening at any other site. This will be determined by assessment of aGVHD response. Acute GVHD will be assessed by Acute GVHD will be assessed by Mount Sinai Acute GVHD International Consortium (MAGIC) algorithm.
Use of High Dose Steroids | Day 28
  The number of subjects requiring high-dose steroids (1mg/kg or greater daily) by Day 28.
Non-relapse mortality. | 6 months
  The number of subjects who expire without relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Sameem Abedin, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No